CLINICAL TRIAL: NCT05005299
Title: The VICTORY Study: A Phase I Study of Venetoclax in Combination With Non-myeloablative Conditioning Allogeneic Haematopoietic Stem Cell Transplantation
Brief Title: Venetoclax in Combination With Non-myeloablative Conditioning Allogeneic Haematopoietic Stem Cell Transplantation
Acronym: VICTORY
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021.238
Record Dates: First submitted 2021-08-08; First posted 2021-08-13 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-06

CONDITIONS: Leukemia, Myeloid, Acute; Leukemia, Lymphoblastic, Acute, L1; Leukemia, Lymphoblastic, Acute, L2; Myelodysplastic Syndromes; Non-hodgkin Lymphoma; Plasma Cell Myeloma
Keywords: Venetoclax; Reduced intensity conditioning; Non-myeloablative conditioning; Allogeneic stem cell transplant; Acute leukemia; Myelodysplastic syndrome; Non-Hodgkin Lymphoma; Plasma Cell Myeloma; Graft-versus-host Disease; Engraftment; Graft-versus-Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Multiple Myeloma; Graft vs Host Disease | interventions — venetoclax; fludarabine; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Phase 1 study, 3+3 design with dose expansion phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose Level A (Experimental): Subjects will receive receive short-course venetoclax on day -11 to -6 [venetoclax 100mg daily administered on day -11 to -6 (total venetoclax dose: 600mg)], followed by intravenous fludarabine 30mg/m2 daily (day -5 to -3) and intravenous cyclophosphamide 750mg/m2 daily (day -5 to -3). Allogeneic stem cell infusion will occur on day 0.
  Interventions: Drug: Venetoclax; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Level B (Experimental): Subjects will receive receive short-course venetoclax on day -11 to -6 [venetoclax 100mg daily administered on day -11, followed by 200mg daily administered on day -10 to -6 (total venetoclax dose: 1100mg)], followed by intravenous fludarabine 30mg/m2 daily (day -5 to -3) and intravenous cyclophosphamide 750mg/m2 daily (day -5 to -3). Allogeneic stem cell infusion will occur on day 0.
  Interventions: Drug: Venetoclax; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Level C (Experimental): Subjects will receive receive short-course venetoclax on day -11 to -6 [venetoclax 100mg daily administered on day -11, followed by 200mg daily administered on day -10, 400mg daily administered on day -9 and 600mg daily administered on day -8 to -6 (total venetoclax dose: 2500mg)], followed by intravenous fludarabine 30mg/m2 daily (day -5 to -3) and intravenous cyclophosphamide 750mg/m2 daily (day -5 to -3). Allogeneic stem cell infusion will occur on day 0.
  Interventions: Drug: Venetoclax; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Level B' (Experimental): Subjects will receive receive short-course venetoclax on day -11 to -6 [venetoclax 100mg daily administered on day -11, followed by 200mg daily administered on day -10 and 400mg daily administered on day -9 to -6 (total venetoclax dose: 1900mg)], followed by intravenous fludarabine 30mg/m2 daily (day -5 to -3) and intravenous cyclophosphamide 750mg/m2 daily (day -5 to -3). Allogeneic stem cell infusion will occur on day 0.
  Interventions: Drug: Venetoclax; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Venetoclax — Venetoclax is administered as an oral tablet once daily.
  Other Names: Venclaxta
Drug: Fludarabine — Fludarabine is administered as an intravenous infusion at a dose of 30mg/m2 daily, to be administered over 30 minutes.
Drug: Cyclophosphamide — Cyclophosphamide is administered as an intravenous infusion at a dose of 750mg/m2 daily, to be administered over 30 minutes and to commence 1 hour after fludarabine infusion.

SUMMARY:
This is a Phase 1, open-label, single center study of short-course oral venetoclax therapy prior to non-myeloablative conditioning with fludarabine and cyclophosphamide in subjects with haematological malignancies who are planned for allogeneic stem cell transplantation (alloSCT). The primary study objective is to determine the safety and maximum tolerated dose of venetoclax when used in combination with fludarabine and cyclophosphamide conditioning. Secondary objectives were to evaluate the transplant outcomes and donor/recipient engraftment of this regimen.

DETAILED DESCRIPTION:
Eligible patients are to be enrolled sequentially into one of 4 treatment Dose Levels (beginning with Dose Level A) to receive short-course venetoclax on day -11 to -6, followed by intravenous fludarabine 30mg/m2 daily (day -5 to -3) and intravenous cyclophosphamide 750mg/m2 daily (day -5 to -3). Allogeneic stem cell infusion will occur on day 0. In the dose-escalation phase of this 3+3 study, three patients are planned for each Dose Level.

Dose Level A: venetoclax 100mg daily administered on day -11 to -6 (total venetoclax dose: 600mg)

Dose Level B: venetoclax 100mg daily administered on day -11, followed by 200mg daily administered on day -10 to -6 (total venetoclax dose: 1100mg)

Dose Level C: venetoclax 100mg daily administered on day -11, followed by 200mg daily administered on day -10, 400mg daily administered on day -9 and 600mg daily administered on day -8 to -6 (total venetoclax dose: 2500mg)

Protocol-specific dose-limiting toxicitues (DLTs) will be assessed from the first dose of venetoclax up to day 30 post-transplant. Subjects will not be treated in a new cohort until all subjects in the previous cohort had completed the DLT evaluation period and ≤ 1 of 6 subjects had experienced a DLT. If ≥ 2 of 6 subjects experienced a DLT at Dose Level C, subjects will be treated at Dose B' as part of the dose-escalation phase of this study.

Dose Level B': venetoclax 100mg daily administered on day -11, followed by 200mg daily administered on day -10 and 400mg daily administered on day -9 to -6 (total venetoclax dose: 1900mg)

The maximum tolerated dose (MTD) is defined as the highest Dose Level at which ≤ 1 of 6 subjects had experienced a DLT. The dose-expansion phase involves recruitment of up to 12 patients at the MTD.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for inclusion if all of the following criteria are met:

* Age ≥ 18 years
* Planned to undergo alloSCT for one of the following haematological malignancies: acute leukaemia (including myeloid and/or lymphoid lineage or biphenotypic), myelodysplastic syndrome, chronic lymphocytic leukaemia (CLL), B-cell non-Hodgkin lymphoma (NHL) and plasma cell myeloma
* Physician preference for a non-myeloablative conditioning regimen
* Available 10/10 HLA-matched related or unrelated haematopoietic stem cell donor
* Transplantation to be performed from a peripheral blood stem cell source
* Adequate renal and hepatic function at screening as follows:

  1. Calculated creatinine clearance >50ml/min as measured by Cockroft Gault formula
  2. AST and ALT ≤ 3.0 x ULN
  3. Bilirubin ≤ 1.5 x ULN (except patients with Gilbert's Syndrome)
* Able to tolerate oral medications
* Disease status at the time of transplantation as follows:

  1. Acute leukaemia in complete morphologic remission
  2. Myelodysplastic syndrome with less than 10% bone marrow blasts
  3. CLL in complete remission (CR), partial response (PR) or PR with lymphocytosis
  4. NHL in CR or PR
  5. Myeloma in CR, very good partial response (VGPR) or PR within 3 months of prior autologous stem cell transplantation as part of a tandem auto-allo transplant approach
* ECOG performance status 0-1

Exclusion Criteria:

Patients will be excluded from this study if any of the following criteria are met:

* Moderate or high risk of tumour lysis syndrome prior to conditioning for allogeneic transplantation, defined as:

  1. For CLL: Diameter of any lymph node or tumour mass >5cm OR absolute lymphocyte count≥25x10^9/L
  2. For NHL: Diameter of any lymph node or tumour mass >5cm
* Prior intolerance of venetoclax or another BCL-2 inhibitor with the exception of cytopenias. Patients with prior clinical tumour lysis syndrome following venetoclax or other BCL-2 inhibitor will be excluded from the study if at the time of prior TLS their disease burden was as follows:

  1. For CLL: Diameter of any lymph node or tumour mass <5cm OR absolute lymphocyte count≤25x10^9/L
  2. For NHL: Diameter of any lymph node or tumour mass <5cm
* Reticulin fibrosis of the marrow of grade MF 2-3
* Prior allogeneic stem cell transplantation
* Haemopoietic cell transplantation - comorbidity index (HCT-CI) score > 5
* Any currently active malignancy other than the primary indication for alloSCT (except localized basal cell carcinoma or squamous cell carcinoma of the skin)
* Uncontrolled systemic infection
* Known malabsorption syndrome
* Has received within 7 days prior to the first dose of venetoclax CYP3A4 inducers such as rifampicin, carbamazepine, phenytoin and St John's wort
* Has received within 7 days prior to the first dose of venetoclax CYP3A4 inhibitors
* Known positivity to HIV
* Significant physical or psychiatric comorbid illness that in the investigator's opinion would impair the patient's ability to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The development of any dose-limiting toxicities | Time point between time of first dose of venetoclax to day 30 post-alloSCT
  Dose-limiting toxicities (DLT), defined as any of the following which cannot be clearly attributed to a concurrent illness, concomitant medication or those expected as part of standard allogeneic stem cell transplant (alloSCT) complications:
  * Any grade 3-4 non-haematological adverse events between day -11 to day -1
  * Primary failure of neutrophil engraftment by day 30 post-alloSCT. The date of neutrophil engraftment is defined as the first of 3 consecutive days of neutrophil count ≥ 0.5 x 10^9/L.
  * Primary failure of platelet engraftment by day 30 post-alloSCT. The date of platelet engraftment is defined as the first day of platelet count ≥ 20 x 10^9/L, with no transfusions for at least 7 days prior.
  * Grade 3-4 acute graft-versus-host disease (GVHD) prior to day 30 post-alloSCT
  * Development of Clinical Tumour Lysis Syndrome

SECONDARY OUTCOMES:
Acute GVHD incidence and severity | 180 days post allo-SCT
  Acute GVHD (grade 1-4 and grade 3-4) is classified according to the Przepiorka criteria
Chronic GVHD incidence and severity | 1-year post-alloSCT
  Chronic GVHD (mild, moderate or severe) is classified according to the Filipovich criteria
GVHD, relapse-free survival (GRFS) incidence | 1-year post-alloSCT
  GRFS is defined as freedom from grade 3-4 acute GVHD, systemic therapy-requiring chronic GVHD, relapse or death in the first year following alloSCT
Relapse and non-relapse mortality incidence | 1-year post-alloSCT
  Relapse is defined as recurrence of disease, determined by radiological or histological grounds.
  Non-relapse mortality is defined as all-cause mortality without recurrence or progressive disease following alloSCT.
Donor/recipient chimerism | Measured at days 30, 60, 100, 1 year and 2 years following alloSCT
  Myeloid and T-cell chimerism by fragment analysis and capillary electrophoresis of shor tandem repeat markers.

CONTACTS AND LOCATIONS:
Overall Officials: David Ritchie, Principal Investigator — Melbourne Health
Locations (1):
- Melbourne Health, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No